CLINICAL TRIAL: NCT03801213
Title: Evaluation of the Bladder Stimulation, a Non-invasive Technique of Urine Collection, in Infant Less Than 6 Months to Diagnose Urinary Tract Infection: a Randomized Multicenter Study
Brief Title: Evaluation of Urine Samples Obtained by Bladder Stimulation for the Diagnosis of Urinary Tract Infection in Infants
Acronym: EEStiVeN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-HPNCL-03
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infection Bacterial
Keywords: Urine Specimen Collection/methods; Infant; Newborn; Feasibility Studies; Bladder stimulation
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinary catheterization (Active Comparator)
  Interventions: Device: urinary catheterization
- manual bladder stimulation Technique (Experimental)
  Interventions: Procedure: manual bladder stimulation technique

INTERVENTIONS:
Device: urinary catheterization — Urinary catheterization with pain controlled
  Arms: Urinary catheterization
Procedure: manual bladder stimulation technique — manual gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 seconds followed by lumbar paravertebral massage maneuvers for 30 seconds. The renal and bladder stimulation will be performed in less than 3 minutes, with a maximum of two attempts spaced about 20 minutes
  Arms: manual bladder stimulation Technique

SUMMARY:
Urinary tract infection (UTI) is the most common serious bacterial infection among infants. Suprapubic aspiration and bladder catheterization are considered as the gold standard by the American Academy of Pediatrics for the diagnosis, yet it is painful and invasive. In contrast, the bladder stimulation technique has been shown to be a quick and non-invasive approach to collect urine in young infants. Actually, the investigators don't have data on bacterial contamination rates for clean-catch midstream urine collections using this technique

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is common in infants and needs to be diagnosed quickly. The risk for urinary tract infection before the age of 2 years is about 1-4% in boys and 3-8% in girls. A delay in diagnosis exposes to severe complications. In infants, the symptoms are not specific. A good urinalysis quality is therefore necessary for the diagnosis of UTI. Different techniques exist to collect urine samples in these children who do not control their urination yet: supra pubic aspiration, catheterization, urine collection bag and clean catch urine. The American Academy of Pediatrics (AAP) recommends supra pubic aspiration (1-9 % bacterial contamination) and urinary catheterization (8-14 % contamination) for collecting urine but these techniques are invasive and painful. The sterile bag is a non-invasive method of urine collection, with a high bacterial contamination rates (26-62%) leading to unnecessary antibiotic treatment. Finally, clean catch urine is an accepted urine sample to diagnose UTI according to the recommendations (13-27 % of bacterial contamination) but this method is only possible for potty-trained children. Recent studies (Herreros et al, Altuntas et al, Tran et al.) have shown that bladder stimulation, which consists of pubic tapping and lumbar massage, would be a new, effective, non-invasive and safe method of collecting urine in infants.

Bladder stimulation may be performed by a nurse or a physician. The steps of the bladder stimulation technique are as follows: (a) cleaning the genital area with warm water and soap b) bladder stimulation technique, requires the presence of 3 people: infants will be held under their armpits by a parent over the bed, with legs dangling in males and hips flexed in females. The nurse or technician will then alternate between bladder stimulation maneuvers: gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 seconds followed by lumbar paravertebral massage maneuvers for 30 seconds. These two stimulation maneuvers will be repeated until micturition begins, or for a maximum of of 3 minutes.

However, the investigators do not have data on the bacterial contamination rate for urine sample using this new technique. the investigators hypothesize that the bladder stimulation is a technique for obtaining urine with a contamination rate equivalent to those obtained by bladder catheterization, in the diagnosis of febrile urinary tract infection in infants under 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants under the age of 6 months
* For whom an urine sample is required for the diagnosis of a urinary tract infection as follows:

  * fever > 39 °C without symptoms
  * fever > 38°C and uropathy or urinary tract infection
  * fever > 38°C and < 3 months
  * fever > 38 °C and > 48h
  * fever > 38 °C with sepsis signs
* Obtaining the authorization of the holders of parental authority
* Affiliation to French social security

Exclusion Criteria:

* Do exhibiting signs of vital distress (respiratory or circulatory or neurological)
* contraindication to bladder catheterization
* antibiotic therapy in the last 48 hours
* antibiotic prophylaxis in the last 48 hours

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Bacterial contamination rates of urine samples per bladder stimulation and urinary catheterization | at 48 hours after inclusion date
  Bacterial contamination of urine sample is defined by:
  * the growth of two or more micro-organisms,
  * or the presence of a non-uropathogenic germ (lactobacilli, Staphylococcus Coagulase negative, Corynebacterium),
  * or a bacteriuria> 0 colony forming unit(CFU)/ml but <104 CFU / ml for bladder catheterization and <105 CFU / ml for clean catch urine collected by bladder stimulation, or leukocyturia <104 / ml

SECONDARY OUTCOMES:
Pain of bladder stimulation | through intervention completion, an average 30 min
  pain is measured by Evaluation ENfant DOuLeur (EVENDOL) scale while the technique is performed. EVENDOL is a pain scale for children under 7. A pain scale validated for children from birth to 7 years. Score ranges from 0 to 15. Treatment threshold: 4/15.
Pain of bladder catheterization | through intervention completion, an average 30 min
  pain is measured by Evaluation ENfant DOuLeur (EVENDOL) scale while the technique is performed. EVENDOL is a pain scale for children under 7. A pain scale validated for children from birth to 7 years. Score ranges from 0 to 15. Treatment threshold: 4/15.
Diagnostic performance of the dipstick urine test | through intervention completion, an average 30 min
  The diagnostic performance of the urinary dipstick will be established through sensitivity , specificity, positive predictive value and negative predictive value taking as Gold Standard cytobacteriological examination of the urine (ECBU). Diagnostic performance, as well as accuracy, will be established in each of the two groups.
  The sensitivity and specificity will be calculated as well as their 95% confidence intervals calculated using the method of the Wilson score
Risk factors associated with the failure of the bladder stimulation technique | through intervention completion, an average 30 min
  for a urinary sample quantity < 2 ml or no urinary sample collected; potential risk factors for failure will be collected (pain, Wight, sex, age, last food and time since las collect urine)

CONTACTS AND LOCATIONS:
Overall Officials: DEMONCHY DIANE, MD, Principal Investigator — Fondation Lenval - Nice Children Hôpitaux Pédiatriques de Nice
Locations (4):
- France (4):
  - CH Antibes Juans les Pins, Antibes
  - CH Grasse, Grasse
  - CHRU Lille, Lille
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice

REFERENCES:
- [Derived] Demonchy D, Ciais C, Fontas E, Berard E, Breaud J, Rohrlich PS, Dubos F, Fortier C, Desmontils J, Herisse AL, Donzeau D, Haas H, Tran A. Evaluation of bladder stimulation as a non-invasive technique for urine collection to diagnose urinary tract infection in infants under 6 months: a randomized multicenter study ("EE-Sti.Ve.N"). Trials. 2019 Dec 27;20(1):783. doi: 10.1186/s13063-019-3914-2. PMID 31881992